CLINICAL TRIAL: NCT05210842
Title: Safety and Efficiency of Electrocautery-enhanced Lumen-apposing Stents - a Single Center Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Antonia Gantschnigg, Principal Investigator, Salzburger Landeskliniken
Other Study IDs: HA Salzburg
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Complication
Keywords: Lumen-apposing metal stents; Complications; Endoscopic ultrasound (EUS)
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumen apposing metal stent: All patients who had a lumen-proximating stent implanted are included.
  Interventions: Other: Endoscopy

INTERVENTIONS:
Other: Endoscopy — The procedures are performed using a flexible therapeutic linear array echoendoscope.

SUMMARY:
Lumen approximating stents have been used in interventional endoscopy to treat retentions in the upper gastrointestinal tract for 10 years. In the last few years, these have also been used with great success to form new anastomoses, especially in palliative patients. In this regard, many studies have been conducted in recent years.

As one of the largest centers for interventional endoscopy in Austria, we have been performing such interventions as standard since 2016.

The use of LAMS has become the standard therapy in many places. Most of the literature describes the technical advantages of LAMS, while the complications are less discussed. Although complications are rare with reported rates below 10%, with the multitude of technological and clinical advances in the field, it is important to understand and manage potential complications such as bleeding, perforation and stent migration.

Our goal is to evaluate the safety, efficacy, and outcome of all EC-LAMS in a single, high-volume center.

Method:

Suitable patients are analyzed retrospectively from the existing database. All patients who had a lumen-proximating stent implanted are included.

DETAILED DESCRIPTION:
Electrocautery-enhanced lumen-apposing stents (EC-LAMS) were originally designed for drainage of the gallbladder, bile duct, and pancreas pseudocysts.

Numerous studies have shown the effectiveness in treating pseudocysts, abscesses and walled-off pancreatic necrosis by creating a cystogastrostomy or cystoenterostomy tract with a LAMS for drainage and necrosectomy.

In patients suffering from acute cholecystitis, unfit for surgery due to significant comorbidities and/or essential need of anticoagulation, percutaneous gallbladder drainage (PTGBD) was considered as the viable treatment option. However, this procedure comes along with a high incidence of complications like bile leak, bowel perforation, catheter displacement, and cholangitis. Several studies compared the outcome of PTGBD with the endoscopic ultrasound-guided gallbladder drainage (EUS-GBD). The results show significantly superior results in the treatment of non-surgical acute cholecystitis patients with EUS-GBD, in order to consider the use of EUS-GBD as the treatment of choice.

Further, newer "off-label indications" of LAMS are to drain the bile duct in case of failed ERCP (endoscopic retrograde cholangiopancreatography) or, in patients where an ERCP is not possible due to malignant distal biliary obstructions, duodenal obstruction, or post-surgery anatomy. The creation of gastro-gastrostomy was used in patients with a gastric bypass to enable to perform an ERCP or drain a postoperative abscess/fluid collection. Results of published studies have already shown satisfactory clinical outcomes in stenting benign structures, mainly strictures near gastrointestinal (GI) anastomoses or due to chronic inflammations (gastroesophageal junction, pylorus).

We aim to evaluate the safety, efficacy, and outcome of all EC-LAMS placed in a single high-volume center.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 99
* Use of an electocautery-assisted lumen apposing stent
* Follow-up of these patients for at least 3 months

Exclusion Criteria:

* Age younger than 18
* No use of an electrocautery-protected lumen-apposing stent
* Lack of follow-up of at least 3 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had a lumen-proximating stent implanted are included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Complications | 2016-2021
  The main outcome measure ist to evaluate how many complications occured during the use of lumen apposing metal stents in a single center

CONTACTS AND LOCATIONS:
Overall Officials: Franz Singhartinger, Dr., Principal Investigator — Salzburger Landeskliniken
Locations (1):
- Salzburger Landeskliniken, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: Undecided